CLINICAL TRIAL: NCT02871427
Title: An Open-label Study of Nelotanserin in Patients With Lewy Body Dementia Who Have Frequent Visual Hallucinations or REM Sleep Behavior Disorder
Brief Title: Open-label Study of Nelotanserin in Lewy Body Dementia With Visual Hallucinations or REM Sleep Behavior Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes to the overall development program for the study medication
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-102-2003
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Lewy Body Dementia; Dementia With Lewy Bodies; Parkinson's Disease Dementia; Visual Hallucinations; REM Sleep Behavior Disorder
Keywords: Lewy body dementia; Dementia with Lewy bodies; Parkinson's disease dementia; Visual hallucinations; REM sleep behavior disorder
MeSH Terms: conditions — Lewy Body Disease; Hallucinations; REM Sleep Behavior Disorder | interventions — nelotanserin

ARMS (1):
- Nelotanserin (Experimental): Once Daily, Oral, at 20, 40, 60, or 80 mg dose
  Interventions: Drug: Nelotanserin

INTERVENTIONS:
Drug: Nelotanserin — Once Daily, Oral, at 20, 40, 60, or 80 mg dose

SUMMARY:
This study seeks to evaluate the long-term safety and effectiveness of nelotanserin for the treatment of visual hallucinations (VHs) and Rapid Eye Movement (REM) Sleep Behavior Disorder (RBD) in subjects with Lewy body dementia (LBD).

DETAILED DESCRIPTION:
This is a multi-center open-label, long-term study in LBD subjects with RBD and/or VHs. Eligible subjects who completed a previous nelotanserin VH or RBD study and choose to participate in this open-label study will receive 20, 40, 60, or 80 mg nelotanserin once daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with LBD who completed a previous nelotanserin VH or RBD study

Exclusion Criteria:

* Subjects with a current serious and/or unstable cardiovascular, respiratory, thyroid, gastrointestinal, renal, hematologic or other medical disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10-20 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability will be evaluated based on incidence of adverse events (AEs) and significant changes in physical examinations, vital signs, ECGs, and clinical laboratory assessments over time during treatment. | 24 weeks
Long-term effectiveness will be evaluated based on change in the frequency and severity of visual hallucinations (as recorded by patient's caregiver) and/or REM sleep behaviors (based on a clinical evaluator) over time during treatment. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences, Inc., Clinical Research
Locations (19):
- United States (19):
  - US120, Birmingham, Alabama
  - US143, Little Rock, Arkansas
  - US114, Boca Raton, Florida
  - US180, Maitland, Florida
  - US154, Ocala, Florida
  - US113, Orlando, Florida
  - US152, Ormond Beach, Florida
  - US107, Indianapolis, Indiana
  - US132, Lenexa, Kansas
  - US103, Rochester, Minnesota
  - US129, Lincoln, Nebraska
  - US101, Chapel Hill, North Carolina
  - US147, Fargo, North Dakota
  - US111, Cincinnati, Ohio
  - US104, Cleveland, Ohio
  - US105, Columbus, Ohio
  - US173, Lincoln, Rhode Island
  - US128, Memphis, Tennessee
  - US131, San Antonio, Texas